CLINICAL TRIAL: NCT01081314
Title: Treating PTSD in Patients With Borderline Personality Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Melanie Harned, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 36517-C; R34MH082143 (NIH)
Record Dates: First submitted 2010-03-03; First posted 2010-03-05 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-11

CONDITIONS: Stress Disorders, Post-Traumatic; Borderline Personality Disorder; Suicide; Self-Injurious Behavior
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Borderline Personality Disorder; Suicide; Self-Injurious Behavior | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard DBT + PTSD Protocol (Experimental): Includes all components of standard DBT (individual therapy, group skills training, phone coaching, and therapist consultation team) plus a modified version of Prolonged Exposure therapy for PTSD.
  Interventions: Behavioral: Dialectical Behavior Therapy; Behavioral: PTSD Protocol
- Standard DBT (Active Comparator): Includes all components of standard DBT (individual therapy, group skills training, phone coaching, and therapist consultation team).
  Interventions: Behavioral: Dialectical Behavior Therapy

INTERVENTIONS:
Behavioral: Dialectical Behavior Therapy — Standard Dialectical Behavior Therapy as described in the 2 DBT treatment manuals (Linehan, 1993a,b).
Behavioral: PTSD Protocol — A modified version of Prolonged Exposure therapy for PTSD
  Arms: Standard DBT + PTSD Protocol

SUMMARY:
Individuals with borderline personality disorder (BPD) are the quintessential multi-problem patients, often presenting to treatment with numerous dysfunctional behaviors and comorbid diagnoses. Dialectical Behavior Therapy (DBT) is a comprehensive, cognitive-behavioral treatment for BPD that has been shown effective in reducing the primary problems it is designed to treat; namely, the frequency and severity of self-injurious and suicidal behavior, maintenance in treatment, and severe problems in living. However, the DBT treatment manual does not currently include a protocol specifying when or how to treat posttraumatic stress disorder (PTSD), a comorbid diagnosis that is prevalent in BPD patients and may maintain or exacerbate BPD criterion behaviors. Similarly, many of the existing treatment outcome studies for PTSD have excluded suicidal, substance abusing, and multiply diagnosed patients, thereby making it difficult to determine the generalizability of these approaches to individuals with BPD. The research proposed here is focused on the development of a protocol based on Prolonged Exposure therapy to treat PTSD in BPD patients that can be integrated into standard DBT, as well as the initial evaluation of this protocol's feasibility, acceptability, and efficacy. The treatment development and pilot testing process will occur in two phases, including measure development and standardization of the treatment protocol via clinical pre-testing (Phase 1); and pilot and feasibility testing of the intervention via a randomized controlled trial (RCT) comparing standard DBT + PTSD Protocol to standard DBT Only (Phase 2). Information gathered during the pilot RCT will be used to inform the design and conduct of a subsequent full-scale RCT. This research has the potential to significantly expand and improve upon the most empirically supported treatment currently available for BPD, while also demonstrating that exposure treatments for PTSD can be implemented safely and effectively in a BPD population.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18-60
* Meet criteria for borderline personality disorder
* Meet criteria for post-traumatic stress disorder
* Can clearly remember at least some part of the traumatic event(s)
* Recent and recurrent self-injurious behavior
* Lives within commuting distance of University of Washington, Seattle campus
* Consents to all research protocols

Exclusion Criteria:

* Male
* Court ordered to treatment
* Diagnosis of psychotic disorder, bipolar disorder, or seizure disorder requiring medication
* Less than 18 years of age or older than 60 years of age
* Problems which by their presence or severity preclude ability to attend or understand treatment and/or requires priority treatment
* Familial or domestic relationship with a current study participant

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2009-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
PTSD Symptom Scale - Interview | Pre-treatment, 4-, 8-, 12-, and 15-months
  A structured clinical interview that measures both the presence and severity of the 17 DSM-IV PTSD symptoms related to specific trauma(s).
Suicide Attempt Self-Injury Interview | Pre-treatment, 4-, 8-, 12-, and 15-months
  A structured clinical interview measuring the topography, intent, medical severity, social context, precipitating and concurrent events, and outcomes of self-injurious and suicidal behavior during a target time period. Each episode is assessed separately and each act is also coded by the assessor (based on all information) as to whether or not it is a suicide attempt.

SECONDARY OUTCOMES:
Treatment History Interview | Pre-treatment, 4-, 8-, 12-, and 15-months
  A structured interview that uses a time-line follow-back method of assessment to describe the participant's involvement with various psychological and medical treatments (e.g., professional psychotherapy, psychiatric hospitalization, physician visits) as well as medications prescribed.
Hamilton Rating Scale for Depression | Pre-treatment, 4-, 8-, 12-, and 15-months
  An interview measuring symptoms of depression.
Dissociative Experiences Scale | Pre-treatment, 4-, 8-, 12-, and 15-months
  A 28-item self-report measure that quantifies the frequency and intensity of a wide range of experiences that are indicative of absorption, dissociation, derealization, amnesia, and depersonalization.
Suicidal Behaviors Questionnaire | Pre-treatment, 4-, 8-, 12-, and 15-months
  A self-report measure of suicide ideation, suicide expectancies, and suicide threats and communications.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie S Harned, Ph.D., Principal Investigator — University of Washington
Locations (1):
- Behavioral Research and Therapy Clinics, University of Washington, Seattle, Washington, United States

REFERENCES:
- [Result] Harned MS, Ruork AK, Liu J, Tkachuck MA. Emotional Activation and Habituation During Imaginal Exposure for PTSD Among Women With Borderline Personality Disorder. J Trauma Stress. 2015 Jun;28(3):253-7. doi: 10.1002/jts.22013. PMID 26062135
- [Result] Harned MS, Korslund KE, Linehan MM. A pilot randomized controlled trial of Dialectical Behavior Therapy with and without the Dialectical Behavior Therapy Prolonged Exposure protocol for suicidal and self-injuring women with borderline personality disorder and PTSD. Behav Res Ther. 2014 Apr;55:7-17. doi: 10.1016/j.brat.2014.01.008. Epub 2014 Feb 11. PMID 24562087
- [Result] Harned MS, Tkachuck MA, Youngberg KA. Treatment preference among suicidal and self-injuring women with borderline personality disorder and PTSD. J Clin Psychol. 2013 Jul;69(7):749-61. doi: 10.1002/jclp.21943. Epub 2013 Feb 26. PMID 23444147
- [Result] Harned MS, Korslund KE, Foa EB, Linehan MM. Treating PTSD in suicidal and self-injuring women with borderline personality disorder: development and preliminary evaluation of a Dialectical Behavior Therapy Prolonged Exposure Protocol. Behav Res Ther. 2012 Jun;50(6):381-6. doi: 10.1016/j.brat.2012.02.011. Epub 2012 Mar 11. PMID 22503959
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Harned MS, Fitzpatrick S, Schmidt SC. Identifying Change Targets for Posttraumatic Stress Disorder Among Suicidal and Self-Injuring Women With Borderline Personality Disorder. J Trauma Stress. 2020 Aug;33(4):610-616. doi: 10.1002/jts.22504. Epub 2020 Mar 26. PMID 32216138
- See also: Behavioral Research and Therapy Clinics — http://depts.washington.edu/brtc/